CLINICAL TRIAL: NCT06296394
Title: Health Outcomes of Parents With Cystic Fibrosis-Aim 2
Acronym: HOPeCF
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Cystic Fibrosis Foundation (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Traci Kazmerski, Assistant Professor, University of Pittsburgh
Other Study IDs: STUDY23080161; 1R01HL161164-01A1 (NIH); KAZMER22A0 (Other Grant/Funding Number: Cystic Fibrosis Foundation)
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Cystic Fibrosis; Parenthood Status
Keywords: cystic fibrosis; parenthood; highly effective modulator therapy
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Parenthood — The intervention group will consist of participants who became first time parents to children under 5 years of age.

SUMMARY:
The goal of this observational prospective study is to determine the health impact of parenthood on United States (US) people with CF in the era of CF transmembrane regulator protein (CFTR) modulators. The investigators will collect physical and mental health data to comprehensively evaluate the impact of parenthood in CF with widespread highly effective CFTR modulator use. The main hypotheses this study aims to examine are:

H1: Parents with CF and moderate-to-severe depression have more rapid change in ppFEV1 (percent predicted forced expiratory volume in one second) versus those with mild or no depression.

H2: Parents with CF who have more parental responsibility and/or stress have more rapid ppFEV1 (percent predicted forced expiratory volume in one second) change than those with less responsibility/stress

H3: Parents using CFTR modulators have decreased ppFEV1 (percent predicted forced expiratory volume in one second) change versus those not using CFTR modulators

Participants will complete quarterly surveys during the first year of parenthood and biannual surveys, thereafter, using the computer-based survey system on an iPad protected for infection control or via personal device or computer via emailed survey link.

DETAILED DESCRIPTION:
The investigators will follow 146 new parents of children <5 years of age at 18 participating US adult CF centers to assess the primary outcome of percent predicted forced expiratory volume in one second (ppFEV1) up to 5 years after becoming a parent. A prospective approach will capture the immediate and long-term impact of the use of the highly effective CFTR modulator ETI (elexacaftor/tezacaftor/ivacaftor) by ~90 percent of US adults with CF. By combining objective health measures and participant surveys, the investigators can comprehensively assess the psychosocial impacts of parenthood and explore the interplay between the parenting role and physical and mental health. The investigators anticipate identifying modifiable factors that may ameliorate negative health impacts of parenthood. The investigators will conduct hypothesis-generating, semi-structured dyadic interviews with a subset of parents and their key supports (partner/family/friend) to inform future interventions. The investigators have selected qualitative methodology to avoid preconceived theories/hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cystic fibrosis via sweat test or genotype analysis
* Became a first-time parent (including foster parent, step parent, adoptive parent, or legal guardian) to a child under 5 years of age within the last 180 days

Exclusion Criteria:

* Undergone a lung transplant
* Does not speak/read English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with cystic fibrosis who have become first-time parents to a child under 5 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2030-02-01 (Estimated); Study Completion 2031-02-01 (Estimated)

PRIMARY OUTCOMES:
Forced Expiratory Volume (FEV1) | Annually from 2 Years prior to enrollment and annually for Year 1 through Year 5
  Rate of change in ppFEV1 as reflected in the medical record from Year 1 to Year 5

SECONDARY OUTCOMES:
Pulmonary Function Tests (PFTs) - Forced Vital Capacity (FVC) | Annually from 2 Years prior to enrollment and annually for Year 1 through Year 5
  Occurrence of PFTs at each clinic visit/hospitalization. Measures include FVC (Forced vital capacity), and the percent predicted.
Pulmonary Function Tests (PFTs) - Forced Expiratory Volume (FEV1) | Annually from 2 Years prior to enrollment and annually for Year 1 through Year 5
  Occurrence of PFTs at each clinic visit/hospitalization. Measures include FEV1(Forced expiratory volume in one second), and the percent predicted.
Pulmonary Function Tests (PFTs) - Forced Expiratory Flow at 25 and 75 percent (FEF25-75) | Annually from 2 Years prior to enrollment and annually for Year 1 through Year 5
  Occurrence of PFTs at each clinic visit/hospitalization. Measures include FEF25-75 (forced expiratory flow at 25 percent and 75 percent of the pulmonary volume), and the percent predicted for each.
History of CF Diagnosis | Year 1
  Date of diagnosis, as reported in the medical record.
History of CF Genotype Information | Year 1
  Genotype information, as reported in the medical record.
History of CF Mutation | Year 1
  Mutation selection, as reported in the medical record.
Number of Hospitalizations | Annually from 2 Years prior to enrollment and annually for Year 1 through Year 5
  The number of hospitalizations, as reported in the medical record, will be used to compute the rate of hospitalizations.
Length of Hospitalizations | Annually from 2 Years prior to enrollment and annually for Year 1 through Year 5
  The length of each hospitalization, as reported in the medical record, will be used to compute the rate of hospitalizations.
Number of Pulmonary Exacerbations | Annually from 2 Years prior to enrollment and annually for Year 1 through Year 5
  The number of pulmonary exacerbations as reported in the medical record will be used to compute the rate of pulmonary exacerbations.
  , hospitalizations (number and length)
Severity of Pulmonary Exacerbations | Annually from 2 Years prior to enrollment and annually for Year 1 through Year 5
  The severity of pulmonary exacerbations (mild, moderate, severe), as reported in the medical record.
Treatment of Pulmonary Exacerbations | Annually from 2 Years prior to enrollment and annually for Year 1 through Year 5
  The type of treatment used for pulmonary exacerbations (IV antibiotic, oral antibiotic), as reported in the medical record.
Rate of Hospitalizations Due to Pulmonary Exacerbations | Annually from 2 Years prior to enrollment and annually for Year 1 through Year 5
  The number and length of hospitalizations, combined, due to pulmonary exacerbations will be used to compute the rate of pulmonary exacerbations.
Clinic Visit Attendance | Annually from 2 Years prior to enrollment and annually for Year 1 through Year 5
  Number of outpatient clinic visits attended, as reported in the Cystic Fibrosis Foundation Patient Registry (CFFPR).
Microbiologic Profile | Annually from 2 Years prior to enrollment and annually for Year 1 through Year 5
  Number of positive screenings of specific types of bacteria, mycobacteria, fungus in cultures as reported in the CFFPR
Medication use | Annually from 2 Years prior to enrollment and annually for Year 1 through Year 5
  Number of positive screenings of medication use, as reported in the medical record, including CFTR modulator therapy, chronic antibiotic use, and home IV treatment.
History of CF-Related Diabetes Status | Annually from 2 Years prior to enrollment and annually for Year 1 through Year 5
  Instances of positive screenings for CF-Related Diabetes as reported in the medical record.
CF-Related Diabetes Control - Hemoglobin A1C | Annually from 2 Years prior to enrollment and annually for Year 1 through Year 5
  Highest Hemoglobin A1C values, as reported in the medical record.
CF-Related Diabetes Control - Glucose Tolerance | Annually from 2 Years prior to enrollment and annually for Year 1 through Year 5
  Oral glucose tolerance test results, as reported in the medical record.
CF-Related Diabetes Control - Insulin Prescription Usage | Annually from 2 Years prior to enrollment and annually for Year 1 through Year 5
  Insulin prescription use and dosage as reported in the medical record
Liver Disease Status | Annually from 2 Years prior to enrollment and annually for Year 1 through Year 5
  Liver disease status (gall stones, liver disease with cirrhosis, liver disease non-cirrhosis, acute liver failure, hepatic steatosis) as reported by the medical record.
Transplantation Status | Annually from 2 Years prior to enrollment and annually for Year 1 through Year 5
  Current transplant status of the patient (not pertinent, accepted on waiting list, evaluated with final decision pending, evaluated and rejected, or had transplantation), as reported in the medical record.
Transplantation Type | Annually from 2 Years prior to enrollment and annually for Year 1 through Year 5
  If participant had transplantation in previous years, the transplant type will also be recorded as shown in the medical record
BMI | Annually from 2 Years prior to enrollment and annually for Year 1 through Year 5
  Height and weight combined, as reported in the medical record, will be collected to calculate BMI and BMI percentile
Sleep Quality | Up to 4 times in Year 1, Up to 2 times in Year 2 through Year 5.
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month period. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Parental Stress | Up to 4 times in Year 1, Up to 2 times in Year 2 through Year 5.
  The Parental Stress Scale is a self-reported questionnaire which assesses feelings and perceptions about the experience of being a parent. Eighteen-item measure with 5-point Likert scale questions from 1 (strongly disagree) to 5 (strongly agree). Score is determined by the sum (possible range of 18 to 90) with higher scores indicating a higher measured level of parental stress.
Life Stressors | Up to 2 times per year in Year 1 through Year 5.
  Holmes-Rahe Life Stress Inventory (HRLSI) is a forty-three-item measure which assesses life stressors by accounting for life events over a 1-year period. Each life event corresponds to a point value (range 11-100). Scores are determined by the sum of the values for all checked life events. Scores of 150 or less refer to a relatively low amount of life change and low susceptibility to stress-induced health breakdowns. Scores of 151 to 300 imply about a 50% chance of a major health breakdown in the next two years. Scores greater than 301 raise the odds of a major health breakdown to about 80%.
Cystic Fibrosis Questionnaire to evaluate quality of life domains | Up to 2 times per year in Year 1 through Year 5.
  The Cystic Fibrosis Questionnaire-Revised (CFQ-R) is a disease-specific instrument designed to measure the impact on overall health, daily life, well-being and symptoms. It consists of 50 individual measures assessing 9 quality of life domains: physical, role/school, vitality, emotion, social, body image, eating, treatment burden, and health perceptions. Each question is scored with the following scales: for questions 1 - 6: Very True = 1, Mostly True = 2, Somewhat True = 3, Not at all True = 4. For questions 7 - 17: Always = 1, Often = 2, Sometimes = 3, Never = 4. For questions 18 - 30: Very True = 1, Mostly True = 2, Somewhat True = 3, Not at all True = 4. For questions 31 - 35: Always = 1, Often = 2, Sometimes = 3, Never = 4. Scaled scores are calculated using the following formula: (Sum of responses - Minimal Possible sum (n x 1)) / (Maximum possible sum (n x 4) - Minimum possible sum (n x 1)) x 100.
Parental Responsibility | Up to 4 times in Year 1, Up to 2 times in Year 2 through Year 5.
  Adapted Parental Responsibility Scale (APRS) is a forty-item measure which assesses responsibility forms of parental involvement. Each form of responsibility is to be rated on a 5-point Likert scale (I always do, I usually do, co-parent and I equally do, co-parent usually does, and co-parent always does) to designate who had primary responsibility for each task.
Daily Care Check-In | Up to 2 times per year in Year 1 through Year 5.
  The Daily Care Check-In Tool is an 18-item measure that assesses the occurrence and frequency of facing barriers to completing treatments over a 6-month period. The Daily Care Check-In Occurrence Scale score can range from 0 (no barriers) to 18 (experiences all barriers). Each barrier is further scored based on a 5-point Likert scale (always, often, sometimes, rarely, never) to assess the frequency of each interference to treatment. Scores for the Daily Care Check-In Interference Scale are calculated by summing the point values assigned to each score. Scores can range from 0 (no barriers) to 90 (experiences all barriers and they always interfere with completing treatments).
Social Support | Up to 4 times in Year 1, Up to 2 times in Year 2 through Year 5.
  Interpersonal Support Evaluation List-Short Form (ISEL-SF) is a 12-item measure that assesses the perceived availability of social support from family, friends, and others. Each statement is scored using a 4-point scale (definitely false, probably false, probably true, definitely true) to measure subscales of appraisal, belonging, and tangible support. All items are summed to a total score ranging from 0 to 36 with higher scores indicating greater perceived social support.
Anxiety | Up to 4 times in Year 1, Up to 2 times in Year 2 through Year 5.
  The Generalized Anxiety Disorder Assessment (GAD-7) is a seven-item measure that is used to assess the severity of generalized anxiety disorder over a 2-week period. The frequency of symptoms is evaluated using a 4-point scale (not at all, several days, more than half the days, nearly every day). The whole scale score can range from 0 to 21. Scores of 0 to 4 indicate minimal anxiety, scores 5-9 indicate mild anxiety, scores 10-15 indicate moderate anxiety and scores greater than 15 indicate severe anxiety.
Depression | Up to 4 times in Year 1, Up to 2 times in Year 2 through Year 5.
  The Patient Health Questionnaire depression scale (PHQ-8) is an 8-item screening tool used to assess depressive symptoms and severity over a 2-week period. The frequency of symptoms is evaluated using a 4-point scale (not at all, several days, more than half the days, nearly every day). Total score (range of 0 to 24) is determined by adding together the scores of each of the items. Scores of 5, 10, 15, and 20 represent the cutoff points for mild, moderate, moderately severe and severe depression, respectively.
Self-Reported Adherence | Up to 2 times per year in Year 1 through Year 5.
  The Self-Reported Adherence to Highly Effective Modulator Therapy scale is a 4-item questionnaire aimed at identifying the class of modulator (ivacaftor, elexacaftor-tezacaftor-ivacaftor, tezacaftor-ivacaftor, lumacaftor-ivacaftor), presence of altered dosing schedules (specific time or days), and missed treatments (yes, no). Adherence is further evaluated by assessing the number of days that treatment occurred as prescribed (0-3 days, 4-6 days, 7-10 days, 11-14 days) over a 2-week period. This measure serves as descriptive data only, and therefore requires no scoring calculations.

CONTACTS AND LOCATIONS:
Overall Officials: Traci M Kazmerski, MD, Principal Investigator — Faculty
Locations (18):
- United States (18):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - National Jewish Health, Denver, Colorado
  - Northwestern University, Evanston, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital/Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of North Carolina, Chapel Hill, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas-Southwestern, Dallas, Texas
  - University of Washington, Seattle, Washington